CLINICAL TRIAL: NCT06992583
Title: Clinical Study of CEA Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) for CEA Positive Advanced Lung Cancer
Brief Title: Targeted Anti-CEA CAR-T Immunotherapy for Advanced Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC089
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced Lung Cancer
Keywords: CEA; CAR-T; Advanced Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted CEA CAR-T intravenous infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T
- Targeting CEA CAR-T pleural infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T

INTERVENTIONS:
Biological: Targeted CEA CAR-T — Subjects meeting the transfusion criteria will receive pre-treatment, which is as follows: fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, and intravenous CEA CAR-T therapy after 1-2 days of rest
  Arms: Targeted CEA CAR-T intravenous infusion group
Biological: Targeted CEA CAR-T — Subjects meeting the reinfusion criteria will receive pre-treatment with fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, rest for 1-2 days, and intraperitoneal reinfusion targeted CEA CAR-T therapy
  Arms: Targeting CEA CAR-T pleural infusion group

SUMMARY:
Lung cancer is the leading cause of morbidity and mortality in the world, of which 80%-85% are non-small cell lung cancer (NSCLC). Most patients with NSCLC are at the advanced stage of diagnosis and have a poor prognosis. The 5-year survival rate of stage III patients is about 15%, the 5-year survival rate of stage IV patients is less than 5%, and the median survival time is only 7 months.

CEACAM5 (CEA), also known as CD66e, is a classic tumor marker that has been used as a marker for many types of tumors for 50 years. It is mainly expressed in lung cancer, esophageal cancer, bile duct cancer, colorectal cancer, gastric cancer and other tumor types.

In previous CAR-T-related clinical trials targeting CEA, the research team found that CAR-T cell preparations had a certain killing effect on CEA positive tumor cells. At the same time, CAR-T cell preparations cannot be sustained for a long time in the body, which is also a key factor restricting the anti-tumor effect of CAR-T cells in the body. To solve this problem, the killing ability and survival ability of CAR-T cell preparations on tumor cells in vitro and in vivo were improved by optimizing CAR structure and improving culture mode.

DETAILED DESCRIPTION:
This study is a single-arm, open, enhanced 3+3 dose-ascending + dose-extending clinical study, aiming to evaluate the safety and efficacy of CAR T cell preparations, initially observe and study the pharmacokinetic characteristics of drugs in CEA positive advanced lung cancer patients, and obtain the recommended dose of CAR T cell preparations for CEA positive advanced lung cancer patients.

Note: The study was initiated on May 8, 2025, with the first participant providing written informed consent on the same date. Due to administrative delays, the registration on ClinicalTrials.gov was completed on May 16, 2025. No study outcomes were accessed, analyzed, or reported prior to the registration. All study procedures strictly adhere to the protocol approved by the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet all of the following criteria to be eligible for enrollment:

1. Age ≥18 years, regardless of gender.
2. Histologically or cytologically confirmed advanced, metastatic, or recurrent lung cancer, including both non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).
3. Disease progression or intolerance after receiving standard therapies (including but not limited to surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy):

   NSCLC: Disease progression or intolerance after at least second-line standard therapy.

   SCLC: Disease progression or intolerance after at least first-line standard therapy.
4. For patients with pleural effusion assigned to the intrapleural infusion group, the pleural effusion volume and characteristics must be accurately assessed by imaging (chest CT or X-ray) combined with cytology. Malignant pleural effusion must be confirmed by the presence of tumor cells in pleural fluid cytology.
5. Tumor CEA positivity confirmed by immunohistochemistry (IHC) within 3 months prior to screening, defined as distinct membranous staining with ≥10% positivity. If the tumor sample was assessed more than 3 months prior to screening, a serum CEA level >10 µg/L is required.
6. At least one measurable lesion according to RECIST 1.1 criteria:

   Non-nodal lesions: longest diameter ≥10 mm. Lymph node lesions: short axis ≥15 mm.
7. ECOG performance status score of 0 to 2 .
8. Estimated life expectancy of more than 12 weeks.
9. No severe psychiatric disorders.
10. Adequate major organ function unless otherwise specified, defined as follows:

    Hematology: WBC > 2.0 × 10⁹/L; Neutrophils > 1.0 × 10⁹/L; Lymphocytes > 0.5 × 10⁹/L; Platelets > 50 × 10⁹/L; Hemoglobin > 80 g/L.

    Cardiac function: LVEF ≥ 50% on echocardiogram; no significant abnormalities on ECG.

    Renal function: Serum creatinine ≤ 2.0 × ULN. Hepatic function: ALT and AST ≤ 3.0 × ULN (≤ 5.0 × ULN if there is hepatic tumor infiltration).

    Total bilirubin ≤ 2.0 × ULN. Peripheral oxygen saturation >92% in room air.
11. Eligible for leukapheresis or venous blood collection, with no contraindications to cell collection.
12. Willing to use reliable and effective contraception methods (excluding rhythm method) from informed consent signing until one year after CAR-T cell infusion.
13. Participant or legally authorized representative has voluntarily signed the informed consent form (ICF), indicating understanding of the study objectives and procedures and willingness to participate in the clinical trial.

Exclusion Criteria:

-

Participants who meet any of the following criteria will be excluded from the study:

1. Clinically symptomatic central nervous system (CNS) metastasis or meningeal metastasis at screening, or other evidence suggesting the presence of uncontrolled CNS or meningeal metastasis, as judged by the investigator.
2. Participation in any other clinical trial within 1 month prior to screening.
3. Vaccination with a live attenuated vaccine within 4 weeks prior to screening.
4. Receipt of the following anti-tumor treatments within 4 weeks prior to screening: chemotherapy, targeted therapy, or any experimental drug treatment within 14 days or at least 5 half-lives (whichever is shorter).
5. Active infection requiring systemic treatment or any uncontrolled infection.
6. Tumor compression of the trachea or major blood vessels, as determined by the investigator to carry a high risk.
7. History of the following cardiac conditions:

   NYHA Class III or IV congestive heart failure. Myocardial infarction or coronary artery bypass graft (CABG) surgery within 6 months prior to enrollment.

   Clinically significant ventricular arrhythmias or a history of unexplained syncope (except due to vasovagal or dehydration-related causes).

   History of severe non-ischemic cardiomyopathy.
8. Active autoimmune disease or any condition requiring long-term immunosuppressive therapy.
9. History of any other untreated malignancy within the past 3 years, except for carcinoma in situ of the cervix or basal cell carcinoma of the skin.
10. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA levels above normal range; positive for hepatitis C antibody with peripheral blood HCV RNA levels above normal range; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis test.
11. Pregnancy or breastfeeding women.
12. Any other condition that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CAR T cell preparations in the treatment of CEA positive advanced lung cancer【safety】 | 28days
  Adverse events and their proportion during the trial (assessed against the Common Terminology Standard for Adverse Events Version 5.0 (CTCAE 5.0) and ASTCT standards)

SECONDARY OUTCOMES:
To evaluate the disease control rate of CAR-T cell preparations in CEA positive advanced lung cancer【efficacy】 | 3months
  Disease control rates at 3 months were assessed according to Response Evaluation Criteria in Solid Tumors,Version 1.1 (RECIST 1.1), including CR, PR, and SD
To evaluate the remission rate of CAR-T cell preparations in CEA positive advanced lung cancer【efficacy】 | 3months
  Objective response rates at 3 months were assessed according to RECIST 1.1, including CR, PR
To evaluate the overall survival of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Overall survival (OS) : The time from the time the subject received CAR T cell retransfusion until death (from any cause)
To evaluate the duration of response of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Duration of response (DOR) : the time from the first evaluation of CR, PR, or SD to the first evaluation of disease recurrence or progression or death from any cause
To evaluate the disease progression-free survival of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Disease progression-free survival (PFS) : the time from the time the subject received CAR T cell therapy until the first disease progression or death from any cause
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Cmax:The highest concentration of CAR T cells amplified in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Tmax:The time to reach the highest concentration of CAR-T cells in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacodynamics】 | 2 years
  The content of free CEA in peripheral blood at each time point after transfusion was determined by immunohistochemical method

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No